CLINICAL TRIAL: NCT01988259
Title: Comparison of Open vs Minimally Invasive Dorsal Approaches for Foraminotomy and Laminoplasty in the Cervical Spine Through Performance of Head-neck-coordination Analysis
Brief Title: Head-neck Coordination Analysis After Minimally Invasive Surgery in the Dorsal Cervical Spine
Acronym: MISDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Schoen Klinik Hamburg Eilbek (Other)
Collaborators: Jacek Cholewicki PhD (Unknown); MSU Center for Orthopedic Research (Unknown)
Responsible Party: Principal Investigator, Ralph Kothe, PD Dr. med., Head of Spine Surgery, Schoen Klinik Hamburg Eilbek
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MISDCS
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Multilevel Cervical Spinal Stenosis; Single Brachial Radiculopathy
MeSH Terms: interventions — Laminoplasty; Foraminotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Bilateral approach for laminoplasty (Active Comparator): Open approach for laminoplasty
  Interventions: Procedure: Bilateral approach for Laminoplasty
- Unilateral approach for laminoplasty (Active Comparator): Minimally invasive approach for laminoplasty
  Interventions: Procedure: Unilateral approach for laminoplasty
- Subperiosteal approach for foraminotomy (Active Comparator): Open approach for foraminotomy
  Interventions: Procedure: Subperiosteal approach for foraminotomy
- Transmuscular approach for foraminotomy (Active Comparator): Minimally invasive approach for foraminotomy
  Interventions: Procedure: Transmuscular approach for foraminotomy

INTERVENTIONS:
Procedure: Bilateral approach for Laminoplasty — Open bilateral approach for laminoplasty in multilevel cervical spinal stenosis
  Arms: Bilateral approach for laminoplasty
Procedure: Unilateral approach for laminoplasty — Unilateral minimally invasive approach for laminoplasty in multilevel cervical spinal stenosis.
  Arms: Unilateral approach for laminoplasty
Procedure: Subperiosteal approach for foraminotomy — Unilateral subperiostal approach for single level foraminotomy
  Arms: Subperiosteal approach for foraminotomy
Procedure: Transmuscular approach for foraminotomy — Unilateral transmuscular approach for single level foraminotomy
  Arms: Transmuscular approach for foraminotomy

SUMMARY:
To proof patients' benefit of minimally invasive surgery in the dorsal cervical spine an apparatus to examine head-neck-coordination was constructed.

Two different surgical techniques will be compared:

Laminoplasty: open approach vs minimally invasive surgery (MIS)-approach; Foraminotomy: open approach vs MIS-approach. Each patient will be tested before surgery, postoperative as well as 3 and 12 month follow-up.

Hypothesis is that patients after MIS-approaches perform better in their head-neck-coordination as patients with open approaches.

ELIGIBILITY:
Inclusion Criteria:

* radicular or myelopathic compression syndrome in the cervical spine

Exclusion Criteria:

* neurological diseases with influence on the neuromuscular function
* previous surgery on the cervical spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Performance of head-neck-coordination after surgery of the dorsal cervical spine | one year
  The primary outcomes of this study are the motor control performance measures assessed using force and position controlled tasks. In addition to motor control performance, secondary outcome measures of patient-oriented outcome measures (e.g. pain, disability, etc.) will be collected.
  Performance measures will consist of the following tasks:
  * Head-Neck Position Tracking - Rotation and Flexion/Extension
  * Head-Neck Force Tracking - Flexion, Extension and Lateral Bending Left/Right
  During the tracking task, a time-varying target (input signal) will be displayed. The participant will be asked to track the specified target by controlling his/her head-neck angle (position tracking) or moment (force tracking). The head position or force during these trials will represent the output signal for the motor control system. These signals will be collected and analyzed in the time and frequency domain to assess error in head-neck motor control.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Kothe, MD, Principal Investigator — Spine Unit @ Schoen Klinik Hamburg Eilbek
Locations (1):
- Schoen Klinik Hamburg Eilbek, Hamburg, Hamburg, Germany